CLINICAL TRIAL: NCT07296757
Title: The Effect of Origami Activities on Comfort Level and Quality of Life in Patients Undergoing Hemodialysis Treatment
Brief Title: The Effect of Origami Activities on Comfort Level and Quality of Life
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Kafkas University (Other)
Responsible Party: Principal Investigator, Helin ATAY, MsC student, Kafkas University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: KAU-SBF-HA-01
Record Dates: First submitted 2025-11-24; First posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Hemodialysis Complication
Keywords: Hemodialysis; Origami; Comfort; Quality of life

STUDY DESIGN:
Intervention Model Description: Experimental: Intervention Group Patients in the intervention group will participate in origami activities three days a week, each lasting approximately 30 minutes.
  No intervention: Control Group Patients in the control group will receive an origami activity booklet and origami paper after the study.
  Each origami activity will be performed using simple shapes, following the order in the researcher-prepared booklet (with the advice of the origami art instructor).
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention (Experimental): group doing origami activities
  Interventions: Other: origami
- Control grup (No Intervention): The group that did not undergo any intervention during hemodialysis and received routine care from nurses

INTERVENTIONS:
Other: origami — origami activity during a hemodialysis session
  Arms: intervention

SUMMARY:
This study was conducted to evaluate the effect of origami activity on the comfort levels and quality of life of patients undergoing HD treatment.

DETAILED DESCRIPTION:
Patients undergoing HD treatment must undergo dialysis 2-3 days a week, spend approximately 4 hours per day at the dialysis center, remain dependent on a center and caregiver throughout the treatment, experience mobility limitations, and experience disruptions in their social relationships. Patients can receive adequate treatment only if their physical, mental, and biochemical well-being are maintained.

Activities implemented by dialysis nurses during hemodialysis can be beneficial for HD patients. Art therapy, which is frequently of interest to individuals (painting, drawing, coloring, mandala painting, mural painting, clay modeling, collage, sculpture, ceramics, and model making), is a therapeutic activity that reduces anxiety, increases awareness, facilitates recovery from trauma, and improves social skills and self-esteem. Its benefits have been proven in various patient groups. Origami art is an art therapy known to provide behavioral, social, emotional, and psychomotor developmental benefits, and its therapeutic effects in HD patients have not been previously studied. In this context, this study aims to make a new scientific contribution to the literature of non-pharmacological nursing interventions by examining the effect of a 12-session origami activity on the comfort level and quality of life of patients undergoing hemodialysis treatment.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older,
* Literate,
* Undergoing continuous hemodialysis treatment for at least six months,
* Receiving hemodialysis treatment three days a week,
* No visual impairment,
* No communication or perception problems and able to communicate in Turkish,
* No issues (wounds, arthritis, orthopedic impairments, etc.) in the upper extremities that would prevent paper folding,
* No arteriovenous fistula in the dominant arm used for folding,
* Has not received a psychiatric diagnosis and is not taking psychiatric medication,
* Voluntarily agrees to participate in the study,
* Has not previously participated in an activity such as origami.

Exclusion Criteria:

* Receiving dialysis treatment as an outpatient,
* Wishing to withdraw from the study at any stage

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-12-08 (Actual); Primary Completion 2026-01-08 (Estimated); Study Completion 2026-01-10 (Estimated)

PRIMARY OUTCOMES:
Hemodialysis Comfort Scale-Version II | Change in comfort at the beginning of the intervention and at the end of the second week and at the end of the fourth week
  Due to the insufficient number of items in the previously developed Hemodialysis Comfort Scale Koşar and colleagues developed the Hemodialysis Comfort Scale -Version II (HDCS-II) scale was developed by Koşar and colleagues, and the same authors conducted validity and reliability studies. The scale consists of 26 items, and the responses to the items are prepared on a five-point Likert scale: never, very rarely, sometimes, very often, always.The scale has six subscales: physical relief, physical relaxation, psychospiritual relaxation, psychospiritual empowerment, environmental empowerment, and sociocultural relaxation. While the scale includes both reverse-scored and forward-scored items, the number of reverse-scored items is predominant. As the score on the scale increases, the patient's comfort also increases.
Kidney Disease Quality of Life Short Form (KDQOLTM-SF 36.1.3) | Change in comfort at the beginning of the intervention and at the end of the fourth week
  The Turkish reliability and validity of the scale developed by Hayy et al. (1994) was established by Yıldırım et al. (2007). The scale consists of 36 items divided into 5 dimensions. These subdimensions are symptom/problem list (12 items), impact of kidney disease (8 items), and burden of kidney disease (4 items). The Likert method is used for scoring each item. Scores range from 0 to 100 in each dimension.

CONTACTS AND LOCATIONS:
Overall Officials: Ayşe Gül Parlak, PhD, Study Director — Kafkas University Health Science Faculty
Locations (1):
- Van Özel Diyaliz Merkezi, Van, Turkey (Türkiye)